CLINICAL TRIAL: NCT00944112
Title: A Feasibility Randomized Trial Comparing Restrictive and Liberal Blood Transfusion Strategies in Patients Requiring Four or More Days in Intensive Care
Brief Title: Restrictive and Liberal Transfusion Strategies in Intensive Care
Acronym: RELIEVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government); Chief Scientist Office of the Scottish Government (Other Government); Transfusion Medicine Education and Research Foundation (Unknown)
Responsible Party: Gemma Watson, The University of Edinburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CZB/4/698; UK Clinical Research Network (Registry Identifier: UKCRN 6606); ISRCTN Register (Registry Identifier: ISRCTN24842715)
Record Dates: First submitted 2009-07-21; First posted 2009-07-23 (Estimated); Last update posted 2011-03-08 (Estimated); Status verified 2011-03

CONDITIONS: Intensive Care; Blood Transfusion; Anemia
Keywords: Intensive care; Blood Transfusion; Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Restrictive RBC Transfusion Group (Experimental): Patients will receive single unit RBC transfusions with a transfusion trigger of ≤70g/L with a target Hb concentration of 71-90g/L during the intervention period.
  Interventions: Biological: Restrictive RBC Transfusion
- Liberal RBC Transfusion Group (Experimental): Patients will receive single unit RBC transfusions with a transfusion trigger of ≤90g/L with a target Hb concentration of 91-110g/L during the intervention period.
  Interventions: Biological: Liberal RBC Transfusion

INTERVENTIONS:
Biological: Restrictive RBC Transfusion — Patients will receive single unit RBC transfusions with a transfusion trigger of ≤70 g/L with a target Hb concentration of 71-90 g/L during the intervention period.
  Other Names: Restrictive Arm
  Arms: Restrictive RBC Transfusion Group
Biological: Liberal RBC Transfusion — Patients will receive single unit RBC transfusions with a transfusion trigger of ≤90 g/L with a target Hb concentration of 91-110 g/L during intervention.
  Other Names: Liberal Arm
  Arms: Liberal RBC Transfusion Group

SUMMARY:
The most effective transfusion practice in critically ill ICU patients is unknown. Currently the data is unclear as to whether a liberal or restrictive transfusion policy is of most benefit to patients in the short and longer term. The aim of this study is to test the hypothesis that liberal use of RBCs (Hb transfusion trigger ≤90g/L; target Hb range 91-110 g/L) to correct anaemia improves clinical outcomes compared with a restrictive transfusion trigger (Hb transfusion trigger ≤70 g/L; target Hb range 71-90 g/L) in anaemic critically ill patients requiring prolonged ICU stay (≥4 days).

Patients will be randomised to one of two transfusion strategies on a 1:1 basis

Group 1 "Restrictive RBC Transfusion group":

Patients will receive single unit RBC transfusions with a transfusion trigger of ≤70 g/L with a target Hb concentration of 71-90 g/L during the intervention period.

Group 2 "Liberal RBC transfusion group":

Patients will receive single unit RBC transfusions with a transfusion trigger of ≤90 g/L with a target of 91-110 g/L during intervention. These patients will all receive a transfusion on the day of randomisation.

Duration of Intervention:

Remainder of ICU stay or 14 days from randomisation, whichever is longer

Follow-Up

Quality of Life, mobility and health service usage questionnaires at 60 and 180 days.

This is a feasibility study that will provide essential data to ensure the success of the full trial. A qualitative study will also be carried out to explore potential reasons for non-recruitment and clinician concerns with the existing protocol. An exploratory biomarker sub-study will test whether a pro-inflammatory signal occurs in the liberally transfused group associated with transfusions.

DETAILED DESCRIPTION:
Anaemia is a common complication of critical illness and 40-50% of all patients in intensive care units (ICUs) receive blood transfusions. However, despite the perceived benefits of correcting anaemia, numerous non-randomised cohort studies and a system review suggest associations between blood transfusions and adverse patient outcomes. The only large randomised controlled trial comparing restrictive with liberal transfusion policies in critically ill patients (the "TRICC study") suggested a trend to greater morality at 30 days in the liberal transfusion group. However the TRICC study does not inform clinical practice with regard to how to manage long stay ICU patients. Also, and importantly, the blood product used in the TRICC study contained white blood cells (non-leucodepleted), which are associated with adverse events, whereas blood in the UK now has the white blood cells removed prior to blood storage (leucodepleted). Due to continuing uncertainty many clinicians continue to use higher Hb transfusion triggers in longer-term ICU patients and we confirmed this recently in a survey of 184 ICU clinicians.

This uncertainty is important for patients, clinicians and the blood services. For example, patients who require longer stays in ICU have long recovery times, use significant hospital resource, and suffer symptoms such as fatigue, breathlessness and reduced Health Related Quality of Life (HRQoL) for many months. It is possible that blood transfusions could alleviate some of these problems. In addition, donated blood is in short supply and is increasingly expensive to produce. As 40% of ICU patients receive transfusions, and use 8% of the Scottish blood stocks, a stronger evidence base could optimise the use of this precious resource.

A Cochrane systematic review (co-authored by one of the applicants, BMcL) noted that current evidence was dominated by the TRICC trial, and concluded that the "....effects of conservative transfusion triggers on functional status, morbidity and mortality, particularly in patients with cardiac disease, need to be tested in further large clinical trials"4. Further studies are clearly required to determine the most effective transfusion practice in critically ill ICU patients.

We have completed an extensive programme of work to inform this study. Based on this data we have identified a patient population in whom an RCT will address many areas of clinical uncertainty. We will study longer-term ICU patients (higher illness severity; higher morbidity; worse long-term functional status; low long-term HRQoL; greater illness costs) who are aged ≥55 (high incidence of IHD; less certainty regarding safety with restrictive approach in TRICC trial). The treatment exposure will last longer than the TRICC trial, potentially including post-ICU care, because anaemia recovers slowly.

This study is a feasibility study comparing the effectiveness of a "restrictive" blood transfusion policy in long-stay ICU patients with a more "liberal" transfusion policy to inform the definitive RCT design. It has been designed to answer the following questions

* What proportion of eligible patients can be recruited to the study?
* What difference in mean Hb concentration and RBCs exposure will occur with our protocol?
* How good is compliance with our proposed study protocol?
* What factors (if any) limit recruitment and result in protocol violations?
* How should the current protocol be modified for a larger definitive trial?
* Are there any strong pro-inflammatory signals or other patient safety concerns associated with liberal RBCs use?
* How should the health economic evaluation be undertaken in the full trial?

This feasibility evaluation includes three elements:

1. A single blind randomised trial comparing patients managed with the restrictive versus the liberal strategy (main study).

2. A comparison of circulating plasma levels of inflammatory biomarkers during the first 24 hours of randomisation in patients managed with the liberal and restrictive strategy.

3. An interview-based qualitative study with clinicians managing patients in the study units.

1. Main Study.

   The overall hypothesis for this programme of work is that liberal use of RBCs to correct anaemia (HB transfusion trigger ≤90g/L; target Hb range 91-110 g/L) improves clinical outcomes compared with a restrictive transfusion trigger (Hb transfusion trigger ≤70g/L; target Hb range 71-90 g/L) in anaemic critically ill patients requiring prolonged ICU stay (≥4 days).

   Patients will be randomised to one of two transfusion strategies on a 1:1 basis

   Group 1 "Restrictive RBC Transfusion group":

   Patients will receive single unit RBC transfusions with a transfusion trigger of ≤70 g/L with a target Hb concentration of 71-90 g/L during the intervention period.

   Group 2 "Liberal RBC transfusion group":

   Patients will receive single unit RBC transfusions with a transfusion trigger of ≤90 g/L with a target of 91-110 g/L during intervention. These patients will all receive a transfusion on the day of randomisation.

   The intervention will last for 14 days from the time of randomisation or until discharge from the intensive care unit, whichever is longer. The aim is for all surviving patients to receive the randomised intervention for at least 14 days in all cases.

   Follow-up Complication rates will be ascertained by case note review during the 60 days following randomisation (hospital stay only).

   The length of their stay in ICU and in hospital will be ascertained from the patient records

   Longer Term follow up of Patients

   Patients will be contacted at 60 and 180 days following randomisation. At these time points the following will be determined or measured:
   * Survival status
   * Physical disability using the Rivermead Mobility Index
   * HRQoL using the SF-12 questionnaire
   * Health economic questionnaire to determine health care resource use (180 days only).
2. Biomarker Study.

   The aim of this part of the study is to explore whether a pro-inflammatory signal is associated with RBC transfusion in intensive care patients. A range of pro- and anti-inflammatory markers will be compared between the patients entering the restrictive group, who are not expected to receive RBCs during the 24 hours following randomisation, and the liberal group, who will all receive at least one RBC unit during the 24 hours following randomisation.

   Blood samples will be collected from patients as follows:

   Restrictive Group: A blood sample will be drawn following randomisation (time zero), at time zero plus 6 hours, and at time zero plus 24 hours.

   Liberal Group: A blood sample will be drawn following randomisation and immediately prior to RBC transfusion (time zero), at time zero plus 6 hours, and at time zero plus 24 hours

   Each blood sample will be 10mL volume (total 30mL per patient). Plasma samples will be batch analysed at the end of the study.
3. Qualitative Study.

The randomised controlled trial (RCT) is widely acknowledged as the "gold standard" in the evaluation of clinical interventions. Recruitment, however, is often problematic, with serious implications for the detection of important treatment differences, the generalisability of research findings to other patient populations and cost. A recent review demonstrated that less than a third of UK studies recruited the required sample size within the timeframe originally specified, and approximately one third required an extended recruitment period. The recruitment and retention of participants is particularly problematic in critical care research, the rationale for which is currently ill-defined.

Review of the existing literature on barriers to research participation suggests that a myriad of methodological/study-specific, organisational and clinician-specific issues exist. The purpose of this exploratory qualitative study, undertaken as part of the RELIEVE programme of work, is to identify and address perceived barriers to recruitment among clinicians prior to a larger definitive trial.

The aims of this study are

* To explore clinicians' experiences of clinical uncertainty in relation to existing guidance (as a default for clinical decision-making) and in relation to recruitment and compliance with the study protocol.
* To explore clinicians' knowledge of and perspectives on existing evidence and guidelines in relation to blood transfusion practice
* To explore clinicians' practice in relation to existing evidence and guidelines
* To explore clinicians' prior perspectives on research participation with particular reference to patient groups (e.g. patients with ischaemic heart disease) or clinical scenarios (e.g. bleeding events) which might elicit clinical uncertainty in relation to recruitment, randomisation or protocol compliance
* To explore clinicians' subsequent experiences of trial participation with reference to previously described concerns
* To develop potential strategies for the improved recruitment and retention of study participants.

Methods We will conduct qualitative semi-structured interviews with clinicians in each of the 6 participating centres. We will invite the Principal Investigator at each site to participate and, in order to minimise selection bias, we will invite a second clinician with a "non-vested interest" in the study to participate. Participants will be interviewed both prior to trial commencement and following trial completion.

Phase I: Prior to study commencement, we will explore (a) clinicians' knowledge and perspectives on existing evidence and guidelines in relation to blood transfusion practice (b) clinicians' practice in relation to existing evidence and guidelines (c) clinicians' perspectives on research participation per se and (d) clinicians' perspectives on the study protocol in relation to patient groups or clinical scenarios which are likely to elicit uncertainty in terms of recruitment, randomisation or protocol adherence.

Phase II: Following study completion, we will invite the same clinicians to describe their experiences and perceptions of trial participation, with particular reference to patient groups or clinical scenarios in which recruitment, randomisation or protocol adherence elicited concern or uncertainty. Using the screening logs, Case Report and Adverse Event Forms kept at each site by the dedicated research nurses, we will explore, where possible, the rationale for (a) clinician refusal of eligible patients and (b) non-compliance with study protocol or (c) withdrawal of recruited patients. We will invite clinicians to identify potential strategies for addressing these issues.

Analysis

The transcribed interviews will be examined and coded for relevant issues using Computer Assisted Qualitative Data Analysis Software (CAQDAS), namely NVIVO8®. Using thematic analysis, we will therefore identify and delineate key issues of concern, as expressed by clinicians, in relation to (a) the recruitment and retention of participants in critical care research (b) the recruitment and retention of eligible patients with reference to the RELIEVE study protocol.

Outcomes

The identification of "generic", protocol-specific and organisational barriers to recruitment will facilitate the identification of clinically and locally relevant strategies to address these issues prior to the larger definitive study. Using both the existing literature and the unique insights provided by this study, we will also develop and refine a screening tool of research barriers which will (a) be used to audit recruitment in the larger definitive study and (b) form the basis of a tool relevant for critical care research per se.

ELIGIBILITY:
Inclusion Criteria:

* The patient remains in the ICU after 96 hours (4 days) or more following ICU admission
* The patient has required mechanical ventilation via an endotracheal tube or tracheostomy tube for 96 hours or more
* The patient is expected to require ≥24 hours of further mechanical ventilation at the time of assessment
* The patient is aged ≥55 years of age
* The patient has a Hb value of 90g/L or less at the time of assessment

Exclusion Criteria:

* Patient with active bleeding at the time of screening
* Patient with traumatic brain injury as presenting diagnosis
* Patient with intracranial haemorrhage as presenting diagnosis
* Patient not expected to survive the next 48 hours at the time of assessment.
* Patient objects to RBC transfusion
* Patient receiving concurrent treatment with erythropoietin or similar erythropoietic agent
* Follow up is not feasible
* Already enrolled in another RCT with similar clinical endpoints

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-08; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Primary outcomes are related to feasibility and include recruitment rate, protocol adherence & difference in mean Hb concentration and RBC exposure between the 2 groups. | 60 days following randomisation

SECONDARY OUTCOMES:
assessment of complication rate in two treatment arms | 60 days following randomisation
assessment of length of stay in ICU and hospital | 60 days following randomisation
Long term follow-up to determine survival status and assess mobility, quality of life & use of health services | 60 and 180 days following randomisation

CONTACTS AND LOCATIONS:
Overall Officials: Timothy S Walsh, MBChB MD MSc, Principal Investigator — NHS Lothian
Locations (6):
- United Kingdom (6):
  - Ninewells Hospital & Medical School, Dundee
  - Royal Infirmary of Edinburgh, Edinburgh
  - Western General Hospital, Edinburgh
  - The Royal London Hospital, London
  - St Thomas' Hospital, London
  - Stirling Royal Infirmary, Stirling

REFERENCES:
- [Background] Marik PE, Corwin HL. Efficacy of red blood cell transfusion in the critically ill: a systematic review of the literature. Crit Care Med. 2008 Sep;36(9):2667-74. doi: 10.1097/CCM.0b013e3181844677. PMID 18679112
- [Background] Hebert PC, Wells G, Blajchman MA, Marshall J, Martin C, Pagliarello G, Tweeddale M, Schweitzer I, Yetisir E. A multicenter, randomized, controlled clinical trial of transfusion requirements in critical care. Transfusion Requirements in Critical Care Investigators, Canadian Critical Care Trials Group. N Engl J Med. 1999 Feb 11;340(6):409-17. doi: 10.1056/NEJM199902113400601. PMID 9971864
- [Background] Walsh TS, Lee RJ, Maciver CR, Garrioch M, Mackirdy F, Binning AR, Cole S, McClelland DB. Anemia during and at discharge from intensive care: the impact of restrictive blood transfusion practice. Intensive Care Med. 2006 Jan;32(1):100-9. doi: 10.1007/s00134-005-2855-2. Epub 2005 Nov 23. PMID 16328221
- [Background] Hill SR, Carless PA, Henry DA, Carson JL, Hebert PC, McClelland DB, Henderson KM. Transfusion thresholds and other strategies for guiding allogeneic red blood cell transfusion. Cochrane Database Syst Rev. 2002;(2):CD002042. doi: 10.1002/14651858.CD002042. PMID 12076437
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Fergusson DA, Pagano MB, Roubinian NH, Turgeon AF, Valentine S, Trivella M, Doree C, Hebert PC. Transfusion thresholds and other strategies for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2025 Oct 20;10(10):CD002042. doi: 10.1002/14651858.CD002042.pub6. PMID 41114449
- [Derived] Radford M, Estcourt LJ, Sirotich E, Pitre T, Britto J, Watson M, Brunskill SJ, Fergusson DA, Doree C, Arnold DM. Restrictive versus liberal red blood cell transfusion strategies for people with haematological malignancies treated with intensive chemotherapy or radiotherapy, or both, with or without haematopoietic stem cell support. Cochrane Database Syst Rev. 2024 May 23;5(5):CD011305. doi: 10.1002/14651858.CD011305.pub3. PMID 38780066
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Trivella M, Roubinian N, Fergusson DA, Triulzi D, Doree C, Hebert PC. Transfusion thresholds for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2021 Dec 21;12(12):CD002042. doi: 10.1002/14651858.CD002042.pub5. PMID 34932836
- [Derived] Jiwaji Z, Nunn KP, Conway-Morris A, Simpson AJ, Wyncoll D, Rossi AG, Walsh TS; RELIEVE Trial Investigators. Leukoreduced blood transfusion does not increase circulating soluble markers of inflammation: a randomized controlled trial. Transfusion. 2014 Oct;54(10):2404-11. doi: 10.1111/trf.12669. Epub 2014 May 5. PMID 24796937
- [Derived] Walsh TS, Boyd JA, Watson D, Hope D, Lewis S, Krishan A, Forbes JF, Ramsay P, Pearse R, Wallis C, Cairns C, Cole S, Wyncoll D; RELIEVE Investigators. Restrictive versus liberal transfusion strategies for older mechanically ventilated critically ill patients: a randomized pilot trial. Crit Care Med. 2013 Oct;41(10):2354-63. doi: 10.1097/CCM.0b013e318291cce4. PMID 23939351
- See also: Edinburgh Clinical Trials Unit website — http://www.clinicaltrials.ed.ac.uk/CurrentTrials.aspx